CLINICAL TRIAL: NCT06173960
Title: 3-year Follow-up of Patients Treated With Jetstream Combined With Ranger for Calcified Femoropopliteal Lesions
Acronym: FIDJI
Status: Completed | Type: Observational
Sponsor: Association de Provence pour la Promotion de l'Enseignement et la Recherche Cardiologique (Other)
Responsible Party: Sponsor
Other Study IDs: FIDJI-2023
Record Dates: First submitted 2023-12-05; First posted 2023-12-18 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Artery Disease
Keywords: Femoropopliteal Lesions
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atherectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with calcified femoropopliteal lesions: Patients presenting calcified femoropopliteal lesions (de novo, unique or multiple, mono or bilateral) and treated by atherectomy with Jetstream combined with Ranger between 1 December 2016 and 31 December 2020
  Interventions: Device: atherectomy

INTERVENTIONS:
Device: atherectomy — Jetstream atherectomy in combination with Ranger paclitaxel elution balloon (Drug Coated Balloon (DCB))

SUMMARY:
The goal of this non interventional study is to evaluate the long-term clinical effects (3-year follow-up after the procedure) of Jetstream atherectomy combined with a paclitaxel-eluting balloon (Ranger) in all patients who were treated for calcified femoropopliteal lesions (de novo, single or multiple, mono- or bilateral) between December 1, 2016 and December 31, 2020 at the Clinique Rhône-Durance, Avignon, France

DETAILED DESCRIPTION:
This study is a non-interventional, retrospective, descriptive, single-centre study of adult male and female patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions, in order to assess the long-term clinical effects of this treatment.

The study will be conducted at the Clinique Rhône-Durance. Data on the management of all adult patients with calcified femoropopliteal lesions treated with Jetstream combined with Ranger between 1 December 2016 and 31 December 2020 will be collected and recorded for analysis.

ELIGIBILITY:
Inclusion Criteria:

* treated for femoropopliteal lesions with Jetstream atherectomy in combination with a Ranger paclitaxel-eluting balloon (Drug Coated Balloon (DCB)) between 1 December 2016 and 31 December 2020.
* Informed and not opposed to the use of their data in this study.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated for femoropopliteal lesions (de novo, single or multiple, mono or bilateral) by Jetstream atherectomy in combination with a Ranger paclitaxel-eluting balloon (Drug Coated Balloon (DCB)) between December 1st, 2016 and December 31st, 2020 at the Rhône-Durance Clinic in Avignon, France, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of the long-term clinical effects (after 3 years of follow-up) of Jetstream atherectomy combined with Ranger - Target Lesion Revascularization | From the date of the procedure until the date of the Target Lesion Revascularization, assessed up to 3 years
  Estimation of median time between the procedure and the Target Lesion Revascularization
Evaluation of the long-term clinical effects (after 3 years of follow-up) of Jetstream atherectomy combined with Ranger - Lesions number and proportion | 3 years after the procedure
  Number and proportion of lesions with absence of Target Lesion Revascularization at 3-year follow-up after the surgery

SECONDARY OUTCOMES:
Evaluation of the 3-year clinical outcome of Jetstream atherectomy combined with Ranger, without reoperation, in patients with calcified femoropopliteal lesions | 3 years following the procedure
  Clinical outcome at 3 years will be assessed by the number and proportion of patients with a reduction in Rutherford category ≥1, or stable at 1 for patients with Rutherford category =1 at inclusion, compared with the baseline value before surgery and without re-intervention
Evaluation of the procedural success of Jetstream atherectomy combined with Ranger in patients with calcified femoropopliteal lesions - stenosis | During the procedure
  The procedural success of Jetstream atherectomy combined with Ranger in patients with calcified femoropopliteal lesions will be assessed at the time of the procedure by the number and proportion of patients with presence of stenosis of residual diameter <30%
Evaluation of the success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions - dissection | During the procedure
  The success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions will be assessed at the time of the procedure by the number and proportion of patients with absence of dissection
Evaluation of the success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions - ruptured vessels | During the procedure
  The success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions will be assessed at the time of the procedure by the number and proportion of patients with presence of ruptured vessels
Evaluation of the success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions - distal embolisation | During the procedure
  The success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions will be assessed at the time of the procedure by the number and proportion of patients with presence of distal embolisation
Evaluation of the success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions - arteriovenous fistula | During the procedure
  The success of the Jetstream atherectomy device combined with Ranger in patients with calcified femoropopliteal lesions will be assessed at the time of the procedure by the number and proportion of patients with presence of arteriovenous (AV) fistula
Assessing the primary patency of Jetstream atherectomy combined with Ranger in patients with calcified femoropopliteal lesions | At 12 months and 36 months
  Primary patency assessed by echo-Doppler
Description of the atherectomy procedure in patients with calcified femoropopliteal lesions - bailout | During the procedure
  Atherectomy procedure described by the number and type of additional stents (bailout) implanted
Description of the atherectomy procedure in patients with calcified femoropopliteal lesions - paclitaxel eluting balloons | During the procedure
  Atherectomy procedure described by the number of paclitaxel eluting balloons, Ranger (Drug Coat Balloons, DCB), used
Check that there is no revascularisation of clinical origin after the surgery - Target Lesion Revascularization | At 1, 6, 12 and 24 months post-procedure
  The absence of revascularisation after the surgery will be verified by the number and proportion of patients with clinically-induced Target Lesion Revascularization
Check that there is no revascularisation of clinical origin after the surgery - Target Vessel Revascularization | At 1, 6, 12, 24 and 36 months post-procedure
  The absence of revascularisation after the surgery will be verified by the number and proportion of patients with clinically-induced Target Vessel Revascularization
Description of the 3-year clinical follow-up of patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions - Rutherford category | At 1, 6, 12, 24 and 36 months post-procedure
  The 3-year clinical follow-up will be described by the number and proportion of patients with an improvement in the Rutherford category (reduction <1) compared with the reference value before surgery
Description of the 3-year clinical follow-up of patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions - Systolic Pressure Index | At 1, 6, 12, 24 and 36 months post-procedure
  The 3-year clinical follow-up will be described by the number and proportion of patients with an improvement in Systolic Pressure Index (SPI) (increase ≥0.10) compared with the baseline value before surgery
Description of the 3-year clinical follow-up of patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions - Deaths | 3 years following the procedure
  The 3-year clinical follow-up will be described by the number and proportion of total deaths and number and proportion of cardiovascular deaths
Description of the 3-year clinical follow-up of patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions - Amputations | At 1, 6, 12, 24 and 36 months post-procedure
  The 3-year clinical follow-up will be described by the number and proportion of patients with major amputations
Description of the 3-year clinical follow-up of patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions - MACE | At 1, 6, 12, 24 and 36 months post-procedure
  The 3-year clinical follow-up will be described by the number and proportion of patients with a major cardiovascular event (MACE)
Description of the 3-year clinical follow-up of patients treated with Jetstream combined with Ranger for calcified femoropopliteal lesions - Repeat surgery | 3 years following the procedure
  The 3-year clinical follow-up will be described by the number and proportion of patients who had a repeat surgery and the total number of repeat surgeries (by cutaneous or bypass route)

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme BRUNET, Dr, Principal Investigator — Clinique Rhône-Durance
Locations (1):
- Clinique Rhône-Durance, Avignon, France